CLINICAL TRIAL: NCT05367622
Title: The Effect of Blood Glucose Monitoring on Behavior Change in Patients With Poorly Controlled Type 2 Diabetes Mellitus
Brief Title: Blood Glucose Monitoring on Behavior Change in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hsiao-Yun Chang, Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ZORPF3M0011
Record Dates: First submitted 2022-04-27; First posted 2022-05-10 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Continuous blood glucose monitoring; Self-regulation; Blood glucose; Diabetes health promotion behavior; Diabetes self-efficacy; Medication compliance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Self-Control; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research investigators and care provider do not participate in the research processes of recruitment, allocation, and intervention. Simple randomization will be assigned subjects into two groups with prepared envelopes in advance. Both groups had intervention, so the participants did not know whether they belonged to the experimental group or the control group. Outcomes assessor and care provider are different persons. Data will be collected according the list of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous glucose monitoring group (Experimental): Self-regulation model of health education will be given for 1-1.5 hrs and telecommunication 10 to 15 minutes for 7 days
  Interventions: Behavioral: Self-regulation health education
- Self-monitoring of blood glucose group (Placebo Comparator): Usual diabetes health education will be given for 1 hr.
  Interventions: Behavioral: Usual diabetes health education

INTERVENTIONS:
Behavioral: Self-regulation health education — 1. Insert the continuous blood glucose monitor
  2. Give self-regulation model of health education to assist patients in making a judgmental decision on how to modify health promotion behaviors to reach a good glucose control
  3. Use Telecommunications on the modifications of health promotion behaviors for 7 days
  Arms: Continuous glucose monitoring group
Behavioral: Usual diabetes health education — 1. Practice self-monitoring of blood glucose
  2. Give usual diabetes health education
  Arms: Self-monitoring of blood glucose group

SUMMARY:
This purpose of this study is to investigate the effect of the self-regulation mode of continuous blood glucose monitoring on blood glucose indicators, self-efficacy, health-promoting behaviors, and medication compliance in patients with Type 2 diabetes. A prospective, randomized, double-blind experimental study is designed with 60 diabetic patients randomly assigned to the experimental group receiving continuous blood glucose monitoring and self-regulation mode of health education and the control group receiving self-monitoring of blood glucose and routine health education. Data will be collected three times, including blood glucose indicators and scales of self-efficacy, health promotion behaviors, and medication compliance.

DETAILED DESCRIPTION:
This purpose of this study is to investigate the effect of the self-regulation mode of continuous blood glucose monitoring on blood glucose indicators, self-efficacy, health-promoting behaviors, and medication compliance in patients with Type 2 diabetes. This study is a prospective, randomized, double-blind experimental study. A total of 60 diabetic patients who are willing to participate in the outpatient clinic of the hospital will be recruited. They are randomly assigned to the experimental group and the control group with 30 patients each. The experimental group will adopt continuous blood glucose monitoring for 7 days and self-regulation mode of health education, while the control group is self-monitoring of blood glucose and routine health education. Data will be collected three times: pre-test, eighth day after intervention, and three-month after intervention. The data included blood glucose indicators and scales of self-efficacy, health promotion behaviors, and medication compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with diabetes by a doctor, and the patient is over 20 years old
2. Hemoglobin A1C (HbA1C)> 8 % or more
3. Possessed self-monitoring equipment for blood glucose
4. ability to use a mobile phone
5. before participation, the subject fully understand the purpose and process of the research and obtain their consent.

Exclusion Criteria:

1. Diabetes health literacy lower than 9 points
2. Those who have difficulty in visual, hearing and speech.
3. Use of diuretics and steroids

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | Pre-test(baseline)
  Blood glucose indicators
Fasting blood glucose | 7 days during intervention
  Blood glucose indicators
Fasting blood glucose | 3 months after intervention
  Blood glucose indicators
24-hr blood glucose | 7 days during intervention
  Blood glucose indicators
HbA1C | Pre-test(baseline)
  Blood glucose indicators
HbA1C | 3 months after intervention
  Blood glucose indicators
Diabetes self-efficacy scale | Pre-test(baseline)
  Use the options of "extremely confident", "moderately confident", "slightly confident" ", "Not very confident", and "Not confident at all" to assess self-efficacy in the performance of diabetes health promotion behaviors; minimum and maximum values are from 17-85 scores, Higher scores mean a better self-efficacy.
Diabetes self-efficacy scale | 8 days after intervention
  Use the options of "extremely confident", "moderately confident", "slightly confident" ", "Not very confident", and "Not confident at all" to assess self-efficacy in the performance of diabetes health promotion behaviors; minimum and maximum values are from 17-85 scores, Higher scores mean a better self-efficacy.
Diabetes self-efficacy scale | 3 months after intervention
  Use the options of "extremely confident", "moderately confident", "slightly confident" ", "Not very confident", and "Not confident at all" to assess self-efficacy in the performance of diabetes health promotion behaviors; minimum and maximum values are from 17-85 scores, Higher scores mean a better self-efficacy.
Diabetes health promoting behavior scale | Pre-test(baseline)
  Use the options of "always", "often", "sometimes", "occasionally", and "never", to assess the performance of diabetes health promotion behaviors; minimum and maximum values are from 17-85 scores, Higher scores mean a better health promoting behaviors.
Diabetes health promoting behavior scale | 8 days after intervention
  Use the options of "always", "often", "sometimes", "occasionally", and "never", to assess the performance of diabetes health promotion behaviors; minimum and maximum values are from 17-85 scores, Higher scores mean a better health promoting behaviors.
Diabetes health promoting behavior scale | 3 months after intervention
  Use the options of "always", "often", "sometimes", "occasionally", and "never", to assess the performance of diabetes health promotion behaviors; minimum and maximum values are from 17-85 scores, Higher scores mean a better health promoting behaviors.
Medication compliance | Pre-test(baseline)
  Use the 5-point Likert scale to assess compliance behaviors; minimum and maximum values are from 0-8 scores, Higher scores mean a wose medication compliance.
Medication compliance | 8 days after intervention
  Use the 5-point Likert scale to assess compliance behaviors; minimum and maximum values are from 0-8 scores, Higher scores mean a wose medication compliance.
Medication compliance | 3 months after intervention
  Use the 5-point Likert scale to assess compliance behaviors; minimum and maximum values are from 0-8 scores, Higher scores mean a wose medication compliance.

SECONDARY OUTCOMES:
Body composition analysis | Pre-test(baseline)
  percentage of fat, bone, and muscle in your body
Body composition analysis | 8 days after intervention
  percentage of fat, bone, and muscle in your body
Body composition analysis | 3 months after intervention
  percentage of fat, bone, and muscle in your body
Diabetes health literacy assessment scale | Pre-test(baseline)
  A person's capacity to obtain, process, and understand basic health information needed to make appropriate health decisions; minimum and maximum values are from 0-12 scores, Higher scores mean a better wose health literacy.
Diabetes health literacy assessment scale | 3 months after intervention
  A person's capacity to obtain, process, and understand basic health information needed to make appropriate health decisions; minimum and maximum values are from 0-12 scores, Higher scores mean a better wose health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- CHENG GUNG MEMORIAL HOSPITAL, Linkou, Taoyuan, Guishan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.